CLINICAL TRIAL: NCT04811209
Title: Determining the Minimum Clinically Important Difference (MCID) and Patient Acceptable Symptom State (PASS) for Acute Pain and Quality of Recovery After Orthopedic Surgery
Brief Title: MCID and PASS for Acute Pain and Quality of Recovery After Orthopedic Surgery
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 20-6059
Record Dates: First submitted 2021-03-17; First posted 2021-03-23 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia | interventions — BCL2-related protein A1; Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- single group, open labelled observational study with no blinding.: All study patients will be managed per routine clinical practice and institutional standard for the performed surgery.
  Interventions: Other: 1.Baseline Measurements Before Surgery; Other: 2.Intraoperative Anesthetic Management; Other: 3.Postoperative Analgesic Management; Other: 4.Postoperative NRS Pain Assessment; Other: 5.Postoperative Global Rating Scale (GRS) Pain Assessment; Other: 6.Postoperative Patient Acceptable Symptom State (PASS) Assessment for Pain; Other: 7.Postoperative Quality of Recovery Assessment; Other: 8.Other Postoperative Assessments

INTERVENTIONS:
Other: 1.Baseline Measurements Before Surgery — * Baseline demographic data
  * Baseline physiological variables (blood pressure, heart rate, respiratory rate, oxygen saturation)
  * Baseline investigations (hemoglobin, coagulation profile, serum electrolytes) if appropriate.
  * Preoperative pain state using NRS (0-10)
  * Preoperative functional state using the QoR-15 questionnaire
  * Pain expectation - patients will be asked preoperatively with the question "In a scale from 0 to 10 (where 0 = no pain and 10 = worst pain imaginable), what do you consider is an acceptable pain score for your first (and second) day after surgery?... Two weeks after surgery?"
  * Pain castastrophizing scale
Other: 2.Intraoperative Anesthetic Management — All study patients will be managed per routine clinical practice and institutional standard for the performed surgery.
Other: 3.Postoperative Analgesic Management — postoperative pain will be managed on the ward using a multimodal analgesic regimen as appropriate. This includes:
  1. acetaminophen 650 - 1,000 mg given orally every 6 hours around the clock
  2. NSAIDs e.g., celecoxib or other agents given orally around the clock per clinical guideline; omit if contraindicated or per surgeon's preference
  3. Opioids e.g., hydromorphone 1-2 mg or oxycodone 15-30 mg given orally every 1-2 hours as required by the patient per standard nurse administered analgesic protocol.
  4. In the event of severe pain refractory to the above treatments, the patient will be offered IV opioid e.g., intermittent doses of 0.2-0.4 mg hydromorphone IV every 10 minutes until pain becomes tolerable
Other: 4.Postoperative NRS Pain Assessment — Pain assessment using NRS pain scores (0 = no pain and 10 = worst possible pain) will be performed by an independent research staff, starting immediately in the PACU and serially over the first 48 hours after surgery or until hospital discharge.
Other: 5.Postoperative Global Rating Scale (GRS) Pain Assessment — Also, the degree of pain relief after treatment is assessed using a subjective 15-point Global Rating Scale (GRS) as mentioned above (Background). This is performed at the same time of each NRS assessment and a minimum of twice daily
Other: 6.Postoperative Patient Acceptable Symptom State (PASS) Assessment for Pain — During each NRS pain assessment before or after an analgesic intervention on POD 0, 1 and 2, the patient will also be asked this question- ""In your opinion, do you consider your current pain state satisfactory after your operation?" Patients giving a positive response are considered having an acceptable pain state. The PASS is the 75th centile for the pain NRS score in those with a satisfactory pain state.
Other: 7.Postoperative Quality of Recovery Assessment — The quality of recovery 15 questionnaire (QoR-15) to measure the dimension of quality of recovery will be administered once in the morning of POD 1 and POD 2. The MCID and PASS for QoR are determined in the same way as for NRS score. The final MCID value will be average of 4 values, 1 generated by the anchor based method and 3 generated by the distribution based method. The PASS for QoR is the 75th centile of the QoR-15 score in those patients who rated their recovery as good.
Other: 8.Other Postoperative Assessments — Additionally, opioid related adverse effects e.g., nausea, vomiting, itchiness, constipation, sedation (RASS + Ramsay)/ and respiratory depression will be assessed daily.

SUMMARY:
This study seeks to define what constitutes an MCID and a PASS in patients undergoing a variety of elective major orthopedic surgery.

DETAILED DESCRIPTION:
Acute postoperative pain after orthopaedic surgery is common and approximately 40% of all surgical patients experience moderate-severe acute postoperative pain. Treatment of acute pain after surgery is important to relieve patient suffering, expedite resumption of activities of daily living, mitigate the risk of postoperative complications, speed ambulation and rehabilitation and hospital discharge. Good pain treatment requires proper and sound pain assessment to guide analgesic therapy. Past studies have determined the MCID values for a variety of chronic pain disorders. There are however limited data on the MCID for acute pain.At the present time, most perioperative acute pain studies use MCID values that are extrapolated from chronic pain studies yet the validity of MCID extrapolation remains unknown. Procedure-specific MCID for pain after most major orthopedic surgery has not been reported.The MCID for a patient reported outcome can be determined using an anchor and a distribution based method.The anchor based method uses a subjective Global Rating Scale (GRS) scale to assess patient's perception of pain relief after treatment. This is a 15-point Likert scale that ranges from -7 to +7 .Another method to determine the MCID value in pain is the distribution based method using mathematical calculations to generate 3 MCID values - 1) 0.3 standard deviation (SD) of mean change in NRS scores, 2) the standard error of measurement (SEM), and 3) 5% of the instrument range of the mean change in the NRS scores after an analgesic intervention according to patient-rated GAR scale. The SEM is calculated as the SD multiplied by the square root of 1 minus the intraclass correlation coefficient. The final MCID value is the average of 4 values, 1 generated from the anchored and 3 generated from the distribution based methods.

The Patient Acceptable Symptom State (PASS) is another measure for patient-reported outcomes. It represents the threshold beyond which patients consider themselves well (satisfied) after an intervention. The PASS is an absolute value, not a change but this value will vary among patients. In essence, PASS indicates a state of wellbeing (feeling good) as opposed to MCID, a state of improvement (feeling better). The 2 concepts are complementary but contrary to MCID, the PASS is the outcome of interest, instead of the extent of improvement. To determine PASS, the patients are asked this question "In your opinion, do you consider your current pain state satisfactory after your operation?" Patients responding "yes" are considered having an acceptable pain state. The PASS is the 75th centile of the pain scale in those who rated their pain state as satisfactory. Higher baseline pain scores are often associated with higher PASS estimates. Little is known about PASS for acute pain after surgery thus a need to determine this benchmark to properly evaluate the clinical benefits of analgesic interventions.

Quality of Recovery (QoR) is another important PRO measure when evaluating the impact of novel intervention strategies. Quality of recovery can be assessed using the QoR-15 questionnaire (scores 0-150) which measures physical & mental well-being as an indication of the quality of recovery after surgery and anaesthesia.

To determine MCID for QoR, both the anchor and distribution based methods will be used. The patient will be asked "How would you rate your overall recovery from surgery since yesterday?" Patients will use the same GRS (-7 to +7) to measure their response. With the anchored-based method, the MCID is the mean change in the QoR-15 score when the patient reports a GRS score of +2 or +3. The distribution-based method will generate 3 other MCID values: 1) 0.3 standard deviation (SD) of the mean change in the QoR score; 2) the standard error of measurement (SEM); and 3) 5% of the instrument range. Again, the final MCID value is the average of 4 values, 1 generated from the anchored and 3 generated from the distribution based methods.

To determine PASS for QoR, the patients will be asked, "In your opinion, have you made a good recovery from your operation?" with response options of yes, no, or unsure. Those who give a positive response is considered having made a good recovery. The PASS for QoR is the 75th centile of the QoR-15 score in those who rated their recovery as good. The only MCID and PASS study by Myles reported a QoR-15 score of 8 & 118 (out of 150), respectively, in patients undergoing a broad range of surgical procedures. Procedure-specific MCID & PASS for QoR-15 after major orthopaedic surgery are currently unknown. Our proposed observational study seeks to define what constitutes an MCID and a PASS in patients undergoing a variety of elective major orthopedic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-80 years
* ASA class I - III
* Primary elective surgery
* unilateral major shoulder surgery e.g., stabilization and arthroplasty procedures:
* unilateral total hip replacement
* unilateral total knee replacement, and
* spinal decompression + fusion involving ≥ 2 levels.
* Hospital admission for ≥ 24 hours after the surgery

Exclusion Criteria:

* Inability to give informed consent
* Poor English comprehension
* Psychiatric disorders e.g., dementia
* Known allergies to morphine / hydromorphone
* Chronic substance abuse and use of recreational drugs
* Any medical disorder that impairs accurate and objective completion of questionnaires

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study patients will be recruited at Toronto Western Hospital
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-06-21 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-11-07 (Estimated)

PRIMARY OUTCOMES:
MCID for NRS pain score after orthopedic surgery | The first 48 hours after 4 types of major orthopedic
  The MCID value represents the change in NRS score after treatment when the patient reports a small improvement of pain relief that corresponds to a GAR score of 2 or 3.

SECONDARY OUTCOMES:
The PASS for NRS pain score after orthopedic surgery | The first 48 hours after 4 types of major orthopedic
  The PASS for NRS pain score after orthopedic surgery
The amount of opioid consumption required to achieve MCID and PASS | The first 48 h hours 4 types of major orthopedic
  The amount of opioid consumption required to achieve MCID and PASS for acute pain after orthopedic surgery.
Quality of recovery | The first 2 days after surgery
  Quality of recovery as assessed using the QoR-15 questionnaire (0-150), higher score means better recovery
The MCID and PASS for QoR-15 | The first 2 days after surgery
  The MCID and PASS for QoR-15 (0-150), higher score means better recovery
The incidence of opioid related adverse reactions and treatments required | The first 2 days after surgery
  The incidence of opioid related adverse reactions and treatments required

CONTACTS AND LOCATIONS:
Overall Officials: Anahi Perlas, MD, FRCPC, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hopspital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No